CLINICAL TRIAL: NCT07337694
Title: Exploring the Clinical Value of an AI-Assisted Patient Self-Assessment App for Bowel Preparation: A Multicenter Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Tianjin Haihe Hospital (Other); Guangdong Second Provincial General Hospital (Other); Dongguan Humen Hospital of Traditional Chinese Medicine (Unknown); Cangzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025ZSLYEC-747
Record Dates: First submitted 2026-01-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Bowel Preparation for Colonoscopy; Colonoscopy
Keywords: Bowel preparation; Colonoscopy; Artificial intelligence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The App group (Experimental): After taking the bowel-prep solution, patients in the app group are instructed to photograph their final stool in the toilet and upload the image through our smartphone app. The AI algorithm immediately scores the prep quality. If the image is rated "poor" or "inadequate," the app displays an alert advising the patient to come to the hospital early or contact clinical staff; clinical staffs then review the photo and decide whether a rescue preparation is needed. The standard rescue was an additional packet of polyethylene glycol. If the image is rated "adequate," the patient is told the prep is acceptable and should proceed to the appointment, where clinical staffs will use the uploaded photo to confirm eligibility for colonoscopy.
  Interventions: Other: The app group
- The control group (No Intervention): The control group followed the conventional procedure: before the examination, clinical staffs asked questions and relied on the patient's verbal description of their stool to judge the adequacy of bowel preparation. If the prep was deemed inadequate, the standard rescue was an additional packet of polyethylene glycol.

INTERVENTIONS:
Other: The app group — After taking the bowel-prep solution, patients in the app group are instructed to photograph their final stool in the toilet and upload the image through our smartphone app. The AI algorithm immediately scores the prep quality. If the image is rated "poor" or "inadequate," the app displays an alert advising the patient to come to the hospital early or contact clinical staff; clinical staffs then review the photo and decide whether a rescue preparation is needed. The standard rescue was an additional packet of polyethylene glycol. If the image is rated "adequate," the patient is told the prep is acceptable and should proceed to the appointment, where clinical staffs will use the uploaded photo to confirm eligibility for colonoscopy.
  Arms: The App group

SUMMARY:
The quality of bowel preparation hinges on how well patients follow the prep-drug regimen, so intensive education is essential. Phone calls, texts, short videos, and mini-programs have all been shown to boost compliance and improve prep quality. Still, we also need a way to spot-early-those patients who are likely to prep poorly so we can step in with a rescue plan.

In our pilot work the investigators built an AI-assisted mini-program that lets patients photograph their effluent and get an instant quality read-out. The single-center RCT showed excellent performance. Because these findings came from one center, the investigators are now launching a multicenter study to test the tool more broadly. Patients will use the AI mini-program at home; if the algorithm predicts inadequate prep it will prompt them to come in early or alert staff so the investigators can initiate a rescue protocol and, ultimately, improve bowel-cleansing quality.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Undergoing colonoscopy at a participating site
3. Able to defecate in a toilet (or in a setting where stool characteristics can be observed) after taking the bowel-prep solution
4. Proficient in using a smartphone
5. Willing to participate voluntarily

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) class III or IV;

  * Gastric-outlet or intestinal obstruction; ③ Active gastrointestinal bleeding; ④ Enterostomy (colostomy/ileostomy); ⑤ Status post total colectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare the bowel preparation quality between the app group and the control group. | Periprocedural
  The rate of adequate and excellent bowel preparation.

SECONDARY OUTCOMES:
Evaluate the diagnostic performance of the app-based assessment. | Periprocedural
  Sensitivity, specificity, negative predictive value, positive predictive value
cecal intubation rate | Periprocedural
cecal intubation time | Periprocedural
withdrawal time (excluding polypectomy and biopsy) | Periprocedural
polyp-detection rate (PDR), adenoma-detection rate (ADR), advanced-adenoma-detection rate (aADR) | Periprocedural
rate of rescue preparation due to inadequate preparation | Periprocedural
clinical staffs' assessment time | Periprocedural
User satisfaction score | Periprocedural
  From 0 to 10, 0 stands for the least satisfaction, and 10 stands for the most satisfaction.
post-procedural adverse events | From enrollment to 30 days after the procedure.
rate of rescheduled examinations due to inadequate preparation | Periprocedural

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-09-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT07337694/Prot_000.pdf
  • Informed Consent Form (2025-12-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT07337694/ICF_001.pdf